CLINICAL TRIAL: NCT00445055
Title: Study of Evaluation of the Profile of Efficiency / Tolerance of 2 Doses of Intravenous Droperidol in the Prevention of the Postoperative Nausea and Vomits Related to the Surgery of the Thyroid
Brief Title: Evaluation of 2 Doses of Intravenous Droperidol in the Prevention of Postoperative Nausea
Acronym: DIPAVO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUBX 2006/02
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Nausea; Vomiting
Keywords: Thyroidectomy; Nausea; Vomiting; Droperidol
MeSH Terms: conditions — Nausea; Vomiting | interventions — Droperidol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Intravenous injection of 0,625 mg Droperidol, 30 min before the end of anesthesia
  Interventions: Drug: Droperidol
- 2 (Experimental): Intravenous injection of 2,5 mg Droperidol, 30 min before the end of anesthesia
  Interventions: Drug: Droperidol
- 3 (Placebo Comparator): Intravenous injection of NaCl 9% (Placebo), 30 min before the end of anesthesia
  Interventions: Drug: Droperidol

INTERVENTIONS:
Drug: Droperidol — Intravenous injection

SUMMARY:
In this prospective, randomised, placebo-controlled study, the researchers determined whether 0.625 mg or 2.5 mg of IV droperidol given 30 min before emergence from general anaesthesia reduces the incidence of immediate and delayed post operative nausea and vomiting (PONV) in thyroid surgical female population. Two hundred and forty six female patients receiving general anaesthesia for thyroid surgery received either droperidol 0.625 mg or droperidol 2.5 mg or placebo before emergence.

DETAILED DESCRIPTION:
* Principal Objective : Our study examined one main question: Are there difference in efficacy between droperidol IV 0.625 mg or 2.5 mg for the treatment or prophylaxis of PONV to surgical patient undergoing thyroid surgery when they receive it 30 min before emergence from general anaesthesia?
* Secondary Objective :

  * comparison of the % of patients in every group:

    * having a complete control of their nausea
    * requiring secondarily the appeal to another anti-emetic treatment in postoperative
    * presenting an Adverse event
  * Compare score of sedation in ach groups
  * Evaluate electrocardiograph
  * Compare the morphine consumption
* Study design : Prospective, randomized, monocenter, double-blind study
* Inclusion criteria :

  * Female
  * More than 18 years old
  * Patients scheduled for thyroid surgery
  * Simplified Apfel score ≥ 2
  * ASA score : 1-2
  * Informed consent obtained from the patient
  * the women in age of procreate must have a reliable contraceptive method
* Exclusion criteria :

  * age < 18 years old
  * male
  * obesity
  * present a severe depressive syndrome
  * pregnancy women
  * trouble of cardiac rate
  * alcoholism
  * contra-indication for Droperidol prescription
* Study plan: three parallel groups will receive 2 different doses of Droperidol or placebo at the end of surgery.

  * Group 1: 0,625mg of Droperidol at the end of surgery
  * Group 2: 2,5mg of Droperidol at the end of surgery
  * Group 3: Placebo at the end of surgery
* Number of subjects : 246

ELIGIBILITY:
Inclusion Criteria:

* Female
* More than 18 years old
* Patients scheduled for thyroid surgery
* Simplified Apfel score ≥ 2
* ASA score : 1-2
* Informed consent obtained from the patient
* Women able to procreate must have a reliable contraceptive method

Exclusion Criteria:

* Age < 18 years old
* Male
* Obesity
* Has a severe depressive syndrome
* Pregnancy women
* Trouble with cardiac rate
* Alcoholism
* Contra-indication for Droperidol prescription

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
No vomiting episode | During the first four hours after intervention

SECONDARY OUTCOMES:
Light nausea | 24h post operative
Control of nausea | 24h post operative
Anti-vomiting treatment | 24h post operative
Adverse events | 24h post operative
Modification of electrocardiograph | 30 min and 120 min after injection
- Score of sedation | 24h post operative

CONTACTS AND LOCATIONS:
Overall Officials: Gérard JANVIER, MD, Study Director — University Hospital, Bordeaux; Laure BAUDOUIN, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Département d'Anesthésie-Réanimation II ; Groupe Hospitalier Sud, CHU de Bordeaux, Pessac, France

REFERENCES:
- [Background] Kovac AL. Prevention and treatment of postoperative nausea and vomiting. Drugs. 2000 Feb;59(2):213-43. doi: 10.2165/00003495-200059020-00005. PMID 10730546
- [Background] Williams OA, Clarke FL, Harris RW, Smith P, Peacock JE. Addition of droperidol to patient-controlled analgesia: effect on nausea and vomiting. Anaesthesia. 1993 Oct;48(10):881-4. doi: 10.1111/j.1365-2044.1993.tb07419.x. PMID 8031342
- [Background] Gan TJ, Meyer T, Apfel CC, Chung F, Davis PJ, Eubanks S, Kovac A, Philip BK, Sessler DI, Temo J, Tramer MR, Watcha M; Department of Anesthesiology, Duke University Medical Center. Consensus guidelines for managing postoperative nausea and vomiting. Anesth Analg. 2003 Jul;97(1):62-71, table of contents. doi: 10.1213/01.ane.0000068580.00245.95. PMID 12818945
- [Background] Wang JJ, Ho ST, Lee SC, Liu YC, Liu YH, Liao YC. The prophylactic effect of dexamethasone on postoperative nausea and vomiting in women undergoing thyroidectomy: a comparison of droperidol with saline. Anesth Analg. 1999 Jul;89(1):200-3. doi: 10.1097/00000539-199907000-00036. PMID 10389804
- [Background] Henzi I, Sonderegger J, Tramer MR. Efficacy, dose-response, and adverse effects of droperidol for prevention of postoperative nausea and vomiting. Can J Anaesth. 2000 Jun;47(6):537-51. doi: 10.1007/BF03018945. PMID 10875717